CLINICAL TRIAL: NCT04559386
Title: Neuromusculaire Monitoring Survey - Usability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EUNeuroMuscMonitoringSurvey3
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-03

CONDITIONS: Survey, Usability
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Participants are asked to fill in a questionnaire and provide extensive information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overall trial (Experimental): People who complete the questionnaire.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Questionnaire

SUMMARY:
This survey aims to better define Anesthesiologist's perceived usability of existing anesthesia Neuromuscular Monitoring devices.

DETAILED DESCRIPTION:
This study consists of a simple online survey that takes approximately 2 minutes to complete.

The study aims to assess Anesthesiologist's perceived usability of the different types of anesthesia neuromuscular monitoring devices (quantitative and qualitative). The survey is targeted to individual anesthesiologists, independetly of their degree of experience.

ELIGIBILITY:
Inclusion Criteria:

* Active Anesthesiology department heads of European Anesthesiology departments.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Usability | 4 months
  Is there a use for Neuromuscular monitoring applications in their department? - questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided